CLINICAL TRIAL: NCT01235806
Title: Contribution of ESAOTE™ Low Field MRI for Diagnosis of Scaphoid Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-CPR-01
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Scaphoid Bone Fracture Suspicion
Keywords: scaphoid; MRI; ESAOTE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI (Other): MRI of the scaphoid bone fracture suspicion
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — MRI of the scaphoid bone fracture suspicion

SUMMARY:
The Alpes Maritimes county administration (France) equipped Nice University Hospital of a 0,2T low field MRI dedicated to distal articulations, devoted to research, installed in the medical imaging unit.

The aim of our project is to study its interest in diagnosis of scaphoid fractures.

Conventional medical care for patients being suspected to have a scaphoid fracture consists in performing a clinical examination and a radiographic check-up with at least 4 incidences, which 2 specific incidences for the scaphoid bone.

Yet, this check up is sometimes defective, causing false positives unnecessary immobilisation and false negatives delays in patient medical care, increasing the risk of complication. Those diagnosis mistakes can bring serious consequences, from permanent partial inability, to professional reclassification.

Alternative imaging exists, but is often irradiating, and never reaches the optimal specificity and sensitivity.

MRI is totally safe, and allows to affirm or invalidate the diagnosis in almost 100% of cases. The problem is the lack of accessibility for emergency cases; therefore there is a great interest in validating the use of a MRI dedicated to distal articulations.

The few studies that study costs of diagnosis strategies including MRI in scaphoid bone fractures diagnosis show a reduction of medical costs if this technique is used early. Our project represents an essential initial step in evaluating the impact of a low field MRI dedicated to peripheral articulations in diagnosis of scaphoid fractures. The next step will be a medico-economical study, since scaphoid fractures occur frequently.

Finally, a new consensus for medical care of scaphoid fracture suspicions could be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of scaphoid bone fracture, whatever the radiologic check-up result is.
* Major patient who signed the informed consent form.
* Patient affiliated to French national health and pensions organization. NON INCLUSION
* MRI contraindication.
* No pain.
* No traumatic antecedent.
* Pregnant or suckler women.
* Patient under a guardianship or a trusteeship
* Patient deprived of liberty consequently to a judiciary procedure
* Patient holding a pace-maker
* Patient holding a foreign body or ferromagnetic prosthetic material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
MRI and radiography interpretation items | The day of the scaphoid fracture
  comparaison between MRI and radiography interpretation items

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas AMORETTI, MD, Principal Investigator — Medical and interventionnal Imaging Unit, Nice University Hospital
Locations (1):
- Medical and Interventionnal Imaging Unit, Archet 2, Nice University Hospital, Nice, France